CLINICAL TRIAL: NCT05330260
Title: Five Years Follow-up of Neurological Outcome After Minimally Invasive Cardiac Surgery: Evidence for Late Cognitive Decline?
Brief Title: Five Years Follow-up of Neurological Outcome After Minimally Invasive Cardiac Surgery
Acronym: FUNOMICS
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Principle Investigator, Jessa Hospital
Other Study IDs: f/2022/012
Record Dates: First submitted 2022-03-03; First posted 2022-04-15 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Surgery; Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Endo-CABG: Group that underwent retrograde arterial cardiopulmonary bypass flow.
  Interventions: Diagnostic Test: neurocognitive test battery
- PCI: Surgical control group
  Interventions: Diagnostic Test: neurocognitive test battery
- Healthy controls: Non-surgical control group
  Interventions: Diagnostic Test: neurocognitive test battery

INTERVENTIONS:
Diagnostic Test: neurocognitive test battery — Assessment of the incidence of late postoperative cognitive decline (LPOCD)

SUMMARY:
A monocenter observational study will be started to investigate postoperative cognitive dysfunction 5 years after minimally invasive cardiac surgery. Postoperative cognitive dysfunction will be evaluated in three groups: an endoscopic-CABG group (endo-CABG), a PCI (Percutaneous Coronary Intervention) group and a healthy control group. It is hypothesized that the endo-CABG group will show a stronger postoperative cognitive dysfunction compared to the PCI group and the healthy control group.

DETAILED DESCRIPTION:
Neurologic complications after cardiac surgery are a major cause of morbidity, prolonged hospital stay and increased costings. In selected cases, postoperative neurologic damage leads to permanent disability or decease of the patient. The American College of Cardiology and the American Heart Association classified neurological sequelae after cardiac surgery into type 1 and type 2. Type 1 morbidities are cardiovascular accident (CVA) and transient ischemic attack (TIA) whereas delirium and postoperative cognitive dysfunction (POCD) are classified as type 2 neurologic injury. Reported incidence of TIA/CVA after coronary artery bypass grafting surgery (CABG) is about 1.6-2%. Incidence of delirium and POCD is more difficult to quantify but ranges from 10-20% for delirium and 30-80% for POCD. Exact pathophysiology remains unclear but seems to be a complex interplay between macro- and microembolization, hypoperfusion and systemic inflammation. Also, preoperative neurologic state might play a role in these frequently comorbid cardiac patients. Some recent papers tried to improve neurologic outcomes by surgical, perfusionist or anesthetic adjustments, with limited success.

Literature concerning neurological complications after minimally invasive cardiac surgery (MICS) is scarce. However, this might be of special concern since in MICS, perfusion to the brain is routinely provided via retrograde flow. By consequence, the brain is possibly exposed to aortic atheroma located distal to the cerebral vessels. This is of special interest since embolic phenomena are identified as a trigger for neurologic failure after cardiac surgery. As the practice of MICS is globally expanding, observations on neurologic outcome after MICS are desirable, with screening for short-term as well as long-term complications.

An important reference article concerning late cognitive outcome after CABG surgery prospectively followed a cohort of 102 CABG patients up until five years after surgery. Patients were tested on eight neurocognitive domains at four moments in time: preoperatively, 3 months after surgery, one year after surgery and ultimately five years after surgery. Somewhat surprisingly, at follow-up on one year after surgery, patients performed significantly better at 5/8 cognitive domains without significant worse scores in the remaining domains. The authors note this finding might be attributed to the learning effect. However, on follow-up after five years, a significant decline in several domains was noted, both compared to one year follow-up as to baseline test results. Unfortunately, due to the lack of a (non-surgical) control group, the authors were unable to attribute this finding to CABG surgery itself or to the normal cognitive evolution in this aging, co-morbid population. Therefore, the group performed a nonrandomized longitudinal prospective study between conventional CABG patients, off-pump CABG (OPCAB) patients, nonsurgical coronary artery patients and healthy controls over a six-year follow-up period. They found a larger decline in all three patient groups compared to the healthy control group although none of the groups was substantially worse compared to baseline. As a result, some authors deduct postoperative neurologic decline is more dependent on preoperative patient state rather influenced by procedure-related factors. However, the influence of MICS and retrograde cardiopulmonary bypass (CPB) flow on long-term neurologic decline remains a question.

Between December 2016 and May 2018 the NOMICS trial (Neurologic Outcome after Minimally Invasive Cardiac Surgery) was performed in Jessa Hospitals, Belgium. Three groups were prospectively followed for three months: an endoscopic-CABG group (endo-CABG), a PCI (Percutaneous Coronary Intervention) group and a healthy age and gender matched control group. A battery of neurocognitive tests was performed in all patients and control group to establish the incidence of POCD. By performing these tests again five years after baseline, the investigators will be able to screen for late cognitive decline in a MICS population undergone retrograde arterial CPB flow. Also, because of the presence of two control groups, it might be able to discriminate if the earlier established late decline is typical to the surgical population, to the coronary artery disease (CAD) population and/or normal aging effect.

ELIGIBILITY:
Inclusion Criteria:

* Minimally 18 years old
* Endo-CABG surgery 5 years ago (group 1)
* PCI surgery 5 years ago (group 2)
* Healthy volunteer 5 years ago (group 3)

Exclusion Criteria:

* Medical history of

  * Stroke or POCD
  * Symptomatic carotid disease
  * Dementia
  * Renal dysfunction (GFR < 30 ml/min)
  * Hepatic dysfunction (Aspartate aminotranspferase (SGOT/AST) or Alanine Amino Transpherase (SGPT/ALT) > 3x normal limits)
* History of drug, medication or alcohol abuse
* Language barrier or inability to communicate
* Physical abnormality that prevents performing the neurocognitive tests
* Surgical revision or presence of intra-operative major cardiac event (endo-CABG)
* Conversion to cardiac surgery of presence of major cardiac event (PCI)
* Simultaneous valve surgery
* Inability to travel to follow-up moment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects that participated in the NOMICS trail 5 years ago were invited to participate in the FUNOMICS trial.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
The incidence of Late postoperative cognitive dysfunction (LPOCD) at 5 years after surgery | through study completion, 5 year follow up after the previous study
  A battery of four tests (Rey Auditory Verbal Learning Test (RAVLT), Trial Making Test (TMT A and B) and the Grooved Pegboard Test) mentioned by the 'statement of consensus on assessment of neurobehavioral outcomes after cardiac surgery', published in 1995 supplemented with two additional tests (ie, the Welscher Adult Intelligence Scale (WAIS)-III digit span test and WAIS-III digit symbol-coding test) will be administered to determine the cognitive outcome. LPOCD is defined as an RCI (Reliable Change Index) ≤-1.645 (significance level 5%) or Z-score ≤-1.645 in at least two different tests.

SECONDARY OUTCOMES:
Comparison of the evolution of LPOCD until five years after the intervention patients (both endo-CABG as PCI) versus five years after baseline for healthy volunteers | through study completion, 5 year follow up after the previous study
  A graph will be created for the group RCI values.
Assessment of predictors of poor neurological outcome after Endo-CABG | through study completion, 5 year follow up after the previous study
  The predictive value of various demographic (ie, age and gender) and perioperative variables on neurological outcome after endo-CABG will be assessed. These variables were already collected for the NOMICS trial.
Assessment of interim medical events: need for additional surgery | through study completion, 5 year follow up after the previous study
  The influence of interim medical events: the need for additional or redo CABG surgery and/or PCI surgery will be assessed.
Quality of life questionnaire | through study completion, 5 year follow up after the previous study
  To compare quality of life (QoL) five years after endo-CABG and PCI the European Quality of Life-5 Dimensions (EQ-5D) questionnaire will be taken. This questionnaire gives a score between 0 and 1 with 1 being the best outcome and 0 being the worst outcome.
Patient satisfaction | through study completion, 5 year follow up after the previous study
  Patient satisfaction five years after endo-CABG and PCI will be assessed with an 11-point numerical rating scale (where 0= not satisfied at all and 10= extremely satisfied).
Interim medical events: brain trauma, dementia, or stroke | through study completion, 5 year follow up after the previous study
  Also formally diagnosed dementia, brain trauma and/or stroke (transient ischemic attack and cerebrovascular accident) will be recorded as interim medical event.
  In line with the 'statement of consensus on assessment of neurobehavioral outcomes after cardiac surgery' a mood state assessment will be performed concurrently. Screening for depression will be performed with the Center for Epidemiological Studies Depression (CES-D) questionnaire.
Interim medical events: depression | through study completion, 5 year follow up after the previous study
  In line with the 'statement of consensus on assessment of neurobehavioral outcomes after cardiac surgery' a mood state assessment will be performed concurrently. Screening for depression will be performed with the Center for Epidemiological Studies Depression (CES-D) questionnaire.
Survival rate 5 years after endo-CABG and PCI | through study completion, 5 year follow up after the previous study

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No